CLINICAL TRIAL: NCT05314140
Title: Towards Optimal Screening and Management of Coronary Artery Disease in Diabetes: TOSCANA Study
Acronym: TOSCANA
Status: Not yet recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Novo Nordisk A/S (Industry); CEBIMER (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-01
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases
Keywords: Coronary artery calcium score; Heart failure risk factors; Prevention; Guidelines
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary artery calcium score evaluation: Patients with diabetes and having a CT scan for evaluation of their coronary artery calcium score will be consecutively include. The indication of the scanner is at the choice of the clinician (usually cardiologist and/or diabetologist), in compliance with the recommendations
  Interventions: Diagnostic Test: Coronary artery calcium score evaluation

INTERVENTIONS:
Diagnostic Test: Coronary artery calcium score evaluation — The evaluation of the coronary artery calcium score will be performed with chest CT scan

SUMMARY:
There are currently only few data on the coronary artery calcium score in patient with diabetes in France, and the diagnostic and therapeutic attitudes towards a high coronary artery calcium score are not standardized and depend on clinical practices, which may vary from one center to another. The proposed multicenter prospective study would provide a better understanding of the epidemiological particularities of the coronary artery calcium score in French diabetics, refine the indications for better performance of the examination, and compare attitudes when this score is high.

DETAILED DESCRIPTION:
The prevalence of coronary heart disease in patient with diabetes varies according to the patient's age, the duration of the diabetes, the coexistence of other heart disease risk factors, but also the type of diagnostic used to detect it. In addition, clinical symptoms are often lacking in diabetic patients.

The latest recommendations from the European Society of Cardiology in 2018 propose a graduation of cardiovascular risk into 3 categories according to the presence of cardiovascular disease, other target organ damage, the duration of diabetes and the coexistence of other heart disease risk factors.

The use of imaging can be considered to refine the cardiovascular risk stratification , such as detection of carotid plaque (class IIa), coronary artery calcium score (class IIb) or even the coronary scanner or ischemia tests (class IIb ). In a much more pragmatic and operational way, the French Society of Cardiology and the Francophone Society of Diabetology very recently published a consensus document, proposing a cardiovascular risk stratification based on clinical elements, the existence of other cardiovascular risk factors and target organ damage risk factors, and the use of the coronary artery calcium score to stratify in particular patients qualified as high risk.

ELIGIBILITY:
Inclusion Criteria:

* Coronary asymptomatic patient
* Patient with type 2 diabetes and aged 50 to 70 or - Patient with type 2 diabetes for more than 10 years and aged 18 to 50 or - Patient with type 1 diabetes for more than 20 years and aged > 35
* Coronary artery calcium score evaluation planned

Exclusion Criteria:

* Patients who already have a clinical history of coronary disease
* Patients with other peripheral arterial disease
* Patients with clinical suspicion of coronary artery disease
* Patients with progressive cancer
* Patients with serious chronic conditions with an estimated life expectancy < 3 years.
* Pregnant, lactating, or pre-menopausal women without a recent negative pregnancy test available.
* Patients under guardianship or curator or placed under justice safeguard
* Patients who do not benefit from the social security scheme, or any equivalent scheme
* Patients refusing or being linguistically or psychologically unable to sign the informed consent form

Participation in another biomedical research protocol is permitted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The centers participating in this study undertake to consecutively include all diabetic patients meeting the selection criteria and having a CT scan for evaluation of coronary artery calcium score. The indication for the scanner is at the choice of the clinician (usually cardiologist and/or diabetologist), in accordance with the recommendations. This is a standard practice study. The patient will be informed of the possibility to participate to the study and his consent will be obtained by the cardiologist/diabetologist when it will be decided to perform a chest CT scan to estimate the coronary artery calcium score. All scanner prescriptions will be carried out according to clinical indications in standard practice.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportions of diabetic patients with high coronary artery calcium score | day 1
  Number of patient with diabetes having a coronary artery calcium score higher than 400

SECONDARY OUTCOMES:
Proportion of patients having a coronary exploration | 6 months
  Number of patient with high coronary artery calcium (>400) score having a coronary exploration compared with patient with low coronary artery calcium score (<400)
Proportion of patients having a myocardial revascularization | 3 months
  Number of patient with high coronary artery calcium score (>400) having a myocardial revascularization compared with patient with low coronary artery calcium score (<400)
Description of adverse events regarding to the coronary artery calcium score | 6 months / 12 months / 18 months / 24 months / 30 months / 36 months / 42 months / 48 months
  Calculation of number and type of cardiovascular adverse event within patient with high coronary artery calcium score (>400) or low coronary artery calcium score (<400)

CONTACTS AND LOCATIONS:
Overall Officials: Victor ABOYANS, MD, Principal Investigator — University Hospital, Limoges; Tessa BERGOT, Study Director — Société Française de la Cardiologie
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Nice, Nice
  - Hôpital Lariboisière, APHP, Paris
  - Hopital Saint Antoine, Paris
  - CHU de Poitiers, Poitiers
  - CHU de la Réunion, Saint-Denis
  - Centre de Cardiologie de Thionville, Thionville
  - CHU de Tours, Tours